CLINICAL TRIAL: NCT04637685
Title: The Enhanse Study The Effect of Infusion Pressure on the Outcomes of Phacoemulsification Surgery
Brief Title: The Effect of Infusion Pressure on the Outcomes of Phacoemulsification Surgery; the ENHANSE Study
Acronym: ENHANSE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: South Tyneside and Sunderland NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 288743
Record Dates: First submitted 2020-10-07; First posted 2020-11-20 (Actual); Last update posted 2020-11-20 (Actual); Status verified 2020-10

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: All outcome assessors will be masked to treatment group allocation. The surgeon will not be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard pressure (Active Comparator): Infusion pressures during phacoemulsification surgeon using the Alcon active sentry system with the Centurion - 70mmHg
  Interventions: Device: Centurion Phacoemulsification System
- Low or physiological pressure (Active Comparator): Infusion pressures during phacoemulsification surgeon using the Alcon active sentry system with the Centurion - 30mmHg
  Interventions: Device: Centurion Phacoemulsification System

INTERVENTIONS:
Device: Centurion Phacoemulsification System — Infusion Pressure

SUMMARY:
The effect of infusion pressure on the outcomes of phacoemulsification surgery.

DETAILED DESCRIPTION:
The Centurion phacoemulsification system with active sentry allows efficient cataract surgery with safe use of high vacuums, whilst allowing low and physiological infusion pressures, significantly lower than other surgical systems. There are reasons to expect that this will lead to patient benefit but it is uncertain if low infusion pressure during phacoemulsification will lead to improved outcomes. This is of particular interest in patients with vascular retinopathies such as diabetic retinopathy where the retinal vasculature is compromised, as well as glaucoma and other optic neuropathies where there is established nerve fibre layer loss.

The investigator will carry out a feasibility study with a two surgeon RCT of 70 patients with diabetic retinopathy and/or glaucoma undergoing phacoemulsification with randomisation of two different infusion pressures (low (30mmHg) versus the higher pressure (~70mmHg) as currently used) using the active sentry system with assessment of a range of exploratory endpoints.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cataract undergoing routine phacoemulsification with either diabetic retinopathy or glaucoma of any degree

Exclusion Criteria:

* Dense cataract precluding adequate retinal imaging
* posterior polar cataract
* subluxated cataract,
* other vision affecting pathology,
* severe glaucoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2021-03-01 (Estimated); Primary Completion 2023-03-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate | From the start to the end of the 10 month planned recruitment period
  The study has been designed as a feasibility study to assess recruitment rate. We will measure rate of recruitment to study (persons per month)

SECONDARY OUTCOMES:
Retinal thickness on SD OCT | Between baseline and day 40
  The above will be measured preoperatively and compared with day 40
Foveal avascular zone size on optical coherence tomography angiography between baseline and day 40 | Between baseline and day 40
  The above will be measured preoperatively and compared with day 40

CONTACTS AND LOCATIONS:
Overall Officials: David Steel, Principal Investigator — South Tyneside and Sunderland NHS Trust

IPD SHARING:
Plan to Share IPD: No